CLINICAL TRIAL: NCT06660433
Title: imProving Respiratory Outbreak Mitigation Through Point-of-care Testing in Long Term Care (PROMPT-LTC): A Cluster Randomized Trial
Brief Title: Respiratory Outbreak Mitigation in Long-Term Care Using Point-of-Care Testing
Acronym: PROMPT-LTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Garron Hospital (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Humber River Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CK-19-2024
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Outbreaks
Keywords: respiratory virus outbreaks; outbreak mitigation; long-term care home

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Point-of-Care Polymerase Chain Reaction Testing Platform (Experimental)
  Interventions: Device: Point-of-care respiratory test platform
- Existing Testing Platform for Respiratory Viruses (Active Comparator)
  Interventions: Other: Existing respiratory virus testing platform

INTERVENTIONS:
Device: Point-of-care respiratory test platform — A point-of-care respiratory multiplex testing platform situated within a long-term care facility to provide rapid test results
  Arms: Point-of-Care Polymerase Chain Reaction Testing Platform
Other: Existing respiratory virus testing platform — Currently used respiratory virus testing platforms
  Arms: Existing Testing Platform for Respiratory Viruses

SUMMARY:
Outbreaks of seasonal respiratory viruses can spread rapidly in long-term care homes. Timely results for diagnostic tests remains a challenge for respiratory viruses due to the logistics of using a reference laboratory with delays leading to missed opportunities to implement virus-specific control measures to interrupt transmission resulting in larger outbreaks. Use of a point-of-care testing platform is a potential solution that provides faster results, but it is uncertain whether this translates into benefits for long-term care residents. This trial aims to assess whether rapid test results for respiratory pathogens (Influenza, Coronavirus disease of 2019 (COVID-19) and Respiratory Syncytial Virus) can impact the number and size of respiratory virus outbreaks in long-term care homes.

ELIGIBILITY:
Inclusion Criteria:

- Long-term care facility engaged with an Ontario Health Team overseen by Sunnybrook Health Science Centre, Michael Garron Hospital or Humber River Health

Exclusion Criteria:

* No signed statement of agreement for study participation
* Pre-existing use of a point-of-care testing platform

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of long-term care residents infected with COVID-19, Influenza, or respiratory syncytial virus (RSV) | 7 months
  The number of long-term care residents who contract Influenza, COVID-19 or RSV separated into the number of residents infected after an introduction is identified and the size of an outbreak of each virus.

SECONDARY OUTCOMES:
The number of outbreaks of Influenza, COVID-19 or RSV | 7 months
  The number of Influenza, COVID-19 or RSV outbreaks as declared by the local Public Health Unit
The number of long-term care residents infected during an outbreak of Influenza, COVID-19 or RSV | 28 days
  The number of long-term care residents with a confirmed or suspected Influenza, COVID-19 or RSV infection during each outbreak as tracked by the local Public Health Unit
Frequency of hospital transfers for long-term care residents infected with Influenza, COVID-19 or RSV | 14 days
  The number of hospital transfers for long-term care residents with Influenza, COVID-19 or RSV
Number of deaths in long-term care residents infected with Influenza, COVID-19 or RSV | 28 days
  The number of long-term care residents who die following an infection with Influenza, COVID-19 or RSV
Duration of outbreaks in of Influenza, COVID-19 or RSV in long-term care facilities | 60 days
  The total duration of an outbreak of Influenza, COVID-19 or RSV as declared by the local Public Health Unit
Secondary attack rate of high-risk exposures to each long-term care resident with Influenza, COVID-19 or RSV infection | 28 days
  The proportion of identified high risk contacts of an infected long-term care resident with Influenza, COVID-19 or RSV infection

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Michael Garron Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan C, Chan CK, Ofner M, O'Brien J, Thomas NR, Callahan J, Pascual B, Palmer SJ, Serapion V, Fabro H, Kozak RA, Candon H, Chan AK, Powis JE, Leis JA. Implementation of point-of-care molecular testing for respiratory viruses in congregate living settings. Infect Control Hosp Epidemiol. 2024 Apr 25;45(9):1-5. doi: 10.1017/ice.2024.72. Online ahead of print. PMID 38659123